CLINICAL TRIAL: NCT00704782
Title: An Open-Label Extension Study of Combination Therapy With Dimebon and Donepezil in Patients With Alzheimer's Disease
Brief Title: Study of Combination Therapy With Dimebon and Donepezil (Aricept) in Patients With Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was halted after a Phase 3 study of dimebon failed to show efficacy.
Sponsor: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIM13
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-11

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — latrepirdine

ARMS (1):
- Dimebon (Experimental): 20 mg by mouth 3 times a day
  Interventions: Drug: dimebon

INTERVENTIONS:
Drug: dimebon

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Dimebon in combination with donepezil (Aricept) in the treatment of Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's disease
* On donepezil (Aricept)
* Caregiver who cares for the patient at least 5 days per week

Exclusion Criteria:

* Unstable medical illnesses or significant hepatic or renal disease
* Other primary psychiatric or neurological disorders

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To assess the safety of Dimebon in combination with donepezil (Aricept) | week 6, 9, 12, 26 and every 13 weeks thereafter until study discontinuation

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Xenoscience, Inc., Phoenix, Arizona
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Barrow Neurological Institute, Phoenix, Arizona
  - Sun Health Research Institute, Sun City, Arizona